CLINICAL TRIAL: NCT05932394
Title: Projection of Visual Material on Postoperative Delirium in Patients Undergoing Cardiac Surgery
Acronym: VisualMaterial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Huelva (Other)
Responsible Party: Principal Investigator, Juan Gómez-Salgado, Professor, University of Huelva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CEIm 2155
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Delirium; Postoperative Delirium; Cardiac Surgery
Keywords: cardiac surgery; delirium; intensive care; visual material; mental health
MeSH Terms: conditions — Delirium; Emergence Delirium; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): In the control group, after the surgical intervention and 30 minutes after the patient's extubation the CAM-ICU scale is administered, recording its value as R0. The following day, at 9:00 a.m., another nurse uses the CAM-ICU scale, noting its value as R1. If postoperative delirium was detected during the day and night, the unit's usual treatment was followed: administration of haloperidol and/or dexmedetomidine.
  Interventions: Behavioral: the usual unit treatment
- Intervention group (Active Comparator): In the intervention group, patients and/or companions are asked to provide visual material, which could consist of photographs of loved ones and/or places known to the patient. 30 minutes after the extubation of the patients, the CAM-ICU scale is administered, recording its value as R0. At night, the projection of images provided by the patient are replaced by a nocturnal visual projection (night sky with stars and moon), ensuring that the patient is able to identify that it was nighttime. Finally, at 9:00 a.m., a nurse who had not worked at night and therefore did not know which patients had received the intervention, administers the CAM-ICU scale again, recording its value as R1.
  Interventions: Behavioral: Projection of Visual Material on Postoperative Delirium in Patients Undergoing Cardiac Surgery

INTERVENTIONS:
Behavioral: Projection of Visual Material on Postoperative Delirium in Patients Undergoing Cardiac Surgery — Patients are randomized into two groups (control group and intervention group). Initially, all patients are administered the "Mini-Mental State Examination scale" (MMSE) to assess their initial cognitive state and their sociodemographic and anthropometric data.
  In the intervention group, patients and/or companions are asked to provide visual material, which could consist of photographs of loved ones and/or places known to the patient. 30 minutes after the extubation of the patients, the CAM-ICU scale is administered.
  In the control group, after the surgical intervention and 30 minutes after the patient's extubation the CAM-ICU scale is administered.
  Arms: Intervention group
Behavioral: the usual unit treatment — CAM-ICU scale is administered to the Control group. No visual material is used.
  Arms: Control group

SUMMARY:
The aim is to evaluate the impact of visual projection of images of relatives or loved ones in patients undergoing cardiac surgery in the immediate postoperative period, and its influence on the incidence and development of postoperative delirium.

A randomized, double-blind clinical trial was designed in the immediate postoperative period of adult patients undergoing cardiac surgery. CONSORT guidelines were followed.

A control group and an intervention group were established. In the intervention group, the patients underwent a visual projection, while the usual unit treatment was carried out with the control group. Sociodemographic, anthropometric, anesthetic, and surgical variables were also recorded. The postoperative delirium assessment scale used was the "Confusion Assessment Method for the Intensive Care Unit scale" (CAM-ICU).

The projection of visual material could reduce the incidence of postoperative delirium in patients undergoing cardiac surgery, although it cannot be established that it is effective as a treatment once the pathology is already established.

The results obtained suggest that the visual projection of images is an effective and economical tool to address an increasingly incidental problem due to the aging of the population.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing heart surgery (aortic valve replacement, mitral valve replacement and/or coronary bypass) in the immediate postoperative period during their stay in the cardiac resuscitation unit.
* Over 18 years of age

Exclusion Criteria:

* Not being sedated for at least 24 hours.
* Leven of consciousness.
* Spanish speaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) scale | 2 times, previous and post intervention, in the first 24 hours after cardiac surgery. This method is applied individually, through study completion, in an average of 1 year.
  Changes in the scale for the diagnosis of delirium in critical care units were assessed previous and post intervention of visual material projection.
  The final CAM-ICU-7 score ranges from 0-7 with 7 being most severe. CAM-ICU-7 scores were further categorized as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Mini-Mental State Examination (MMSE) scale | Baseline (Beginning of the experiment)
  Initially, regardless of the group to which they belonged, all patients were administered the MMSE scale to assess their initial cognitive state and their sociodemographic and anthropometric data were collected.
  The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Leon, León, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data available under reasonable request to the principal investigator.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT05932394/SAP_000.pdf